CLINICAL TRIAL: NCT03158662
Title: Survey to Identify Burdens and Unmet Needs of EB Patients in the US
Brief Title: Survey to Identify Burdens and Unmet Needs of Patients With Epidermolysis Bullosa
Status: Completed | Type: Observational
Sponsor: Amicus Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: EB Survery 2017
Record Dates: First submitted 2017-05-10; First posted 2017-05-18 (Actual); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Epidermolysis Bullosa
Keywords: Epidermolysis Bullosa; Recessive Dystrophic; Simplex; Junctional Non-Herlitz
MeSH Terms: conditions — Epidermolysis Bullosa | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — Survey Study

SUMMARY:
This survey intends to collect information on key aspects of life with epidermolysis bullosa (EB), including diagnostic journey, treatment, management, daily living challenges, and overall psycho-social, socio-economic, academic and family impact.

Objectives:

* To understand the unmet needs for people living with EB in the US
* To assess the differences/similarities in the management/treatment of EB patients (including wound care, symptom management and other issues)
* To assess the EB patients' and caregivers' perceptions of current management/treatment
* To assess the challenges and the burden of daily living with EB
* To understand EB diagnostic journey (the time to diagnosis and by what type of healthcare provider)
* To identify professional disciplines involved in the diagnosis and management of EB
* To understand the psycho-social, socio-economic, academic, and family impact of EB

DETAILED DESCRIPTION:
Epidermolysis bullosa (EB) is a rare, often severe genetic disorder characterized by mechanical fragility and blistering or erosion of the skin, mucosa, or epithelial lining of other organs, in response to little or no apparent trauma.

EB is chronic, potentially disfiguring, and in some cases fatal. Patients with EB have painful wounds and blisters that can lead to infection and scarring. There are many genetic and symptomatic variations of EB, but all forms share the common symptom of fragile skin that blisters and tears, sometimes from the slightest friction or trauma. There is currently no approved treatment for EB. Current standard of care consists of pain management and the bandaging and cleaning of open wounds to prevent infection.

While there are a number of publications/guidance/consensus statements related to the diagnosis and management of EB from the point of view of the health-care provider/disease expert, there is a need for more research to define the key aspects of life with EB (i.e. diagnostic journey, treatment, management, daily living challenges, and overall disease burden) from the perspective of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of EB including subtype
* Resident of the US
* Informed Consent
* Patient must be 18 years or older
* If the survey is done by a caregiver, they must be a parent or legal guardian and must be 18 years or older to answer on behalf of a patient under 18 years or on behalf of a patient 18 years or older who is unable to answer for themselves.
* Must participate in and complete a one hour telephone interview

Exclusion Criteria:

* Patient failing to meet the inclusion criteria above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: EB Patients 18 years of age or older or caregivers of patients under 18 years of age
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2017-04-02 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Current quality of life burdens for EB patients | Outcome will be assessed immediately after subjects answer the questionnaire as this is a cross-sectional survey

CONTACTS AND LOCATIONS:
Locations (1):
- Amicus Therapeutics, Cranbury, New Jersey, United States